CLINICAL TRIAL: NCT07262671
Title: Exosome Detection for Predicting Treatment Efficacy in Advanced NSCLC With Malignant Pleural Effusion
Brief Title: Predictive Value of Exosomes in Pleural Effusion for Advanced Lung Cancer
Acronym: MPE-NSCLC
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Professor, Fudan University
Other Study IDs: MPE-NSCLC-2025
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The following types of biospecimens will be collected and retained for research purposes in this study:
  Peripheral Blood: Approximately 8 mL of venous blood will be collected in EDTA anticoagulant tubes.
  Malignant Pleural Effusion (MPE): Approximately 4 mL of freshly drained pleural fluid will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC-MPE: advanced NSCLC with Malignant Pleural Effusion

SUMMARY:
The goal of this observational study is to investigate the predictive value of exosome characteristics in patients with advanced non-small cell lung cancer (NSCLC) and malignant pleural effusion (MPE). The main question it aims to answer is:

Can the long RNA profile of exosomes derived from plasma and malignant pleural effusion predict treatment response in patients with advanced NSCLC and MPE? Participants who are scheduled to receive standard systemic therapy (including immunotherapy, chemotherapy, or targeted therapy) as part of their regular medical care will be enrolled. Researchers will collect paired samples of peripheral blood and malignant pleural effusion at baseline and key time points during treatment to analyze the exosomal long RNA profiles and correlate them with treatment efficacy and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Confirmed advanced-NSCLC Aged 18-75 years. ECOG performance status of 0-1. At least one measurable lesion as per RECIST 1.1. Adequate bone marrow, liver, and renal function. Willing and able to provide written informed consent.

Exclusion Criteria:

- Mixed small cell lung cancer histology. Symptomatic or untreated brain metastases. Uncontrolled cardiovascular diseases or severe comorbidities. Active hepatitis B/C or HIV infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll approximately 100-120 patients with histologically or cytologically confirmed stage IV NSCLC who present with MPE and are scheduled to receive standard systemic therapy (including but not limited to immunotherapy, chemotherapy, or targeted therapy).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-10-16 (Estimated); Study Completion 2030-10-16 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | From date of enrollment until the first documented progression or death from any cause, assessed up to 24 months.
  Primary Objective: To investigate the association between baseline exLR expression profiles in plasma and malignant pleural effusion and the objective response rate (ORR) as assessed by RECIST 1.1 in patients with advanced NSCLC and MPE receiving systemic therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jialei Wang, MD, Principal Investigator — Shanghai Cancer hospital Fudan University
Locations (1):
- Shanghai Cancer hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes